CLINICAL TRIAL: NCT02585791
Title: EVALUATION OF ACUTE AND SUBACUTE EFFECTS OF NICOTINE FREE ELECTRONIC CIGARETTE (NFEC) VAPORS -Aim 2.1 of "Adverse Effects of Inhaled Nicotine From Tobacco and E-cigarettes".
Brief Title: Evaluation of Acute and Subacute Effects of Nicotine Free Electronic Cigarette(NCFE) Vapors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to recent release reports from CDC about lung injury due to vaping, the PI and IRB decided to terminate the study
Sponsor: University of Miami (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Principal Investigator, Michael Campos, MD, Associate Professor, University of Miami
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 20150373
Record Dates: First submitted 2015-10-22; First posted 2015-10-23 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Healthy Lifetime Non-smokers
Keywords: electronic cigarette; airway inflammation; nasal potential difference
MeSH Terms: conditions — Vaping | interventions — Propylene Glycol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- vape NFEC containing 100% PG (Experimental): Subjects will then be instructed how to use the NFEC (eGo-T® with light emitting diode (LED) display) for 1 week of regularly vaping NFEC containing 100% Propylene Glycol . Subjects will be given the eGo-T®, which contains a 1.2 ml refillable cartridge and a 1100 mAh battery with an LED display to record the number of puffs. Subjects will be asked to puff 100x per day (equivalent to ~10-11 cigarettes) for 7 days. We will accept a vaping range of 80-120 times a day.
  Interventions: Other: Propylene Glycol
- vape 100% vegetable glycerin -VG (Experimental): Subjects will then be instructed how to use the NFEC (eGo-T® with LED display) for 1 week of regularly vaping NFEC containing 100% VG. Subjects will be given the eGo-T®, which contains a 1.2 ml refillable cartridge and a 1100 mAh battery with an LED display to record the number of puffs. Subjects will be asked to puff 100x per day (equivalent to ~10-11 cigarettes) for 7 days. We will accept a vaping range of 80-120 times a day.
  Interventions: Other: vegetable glycerin
- vape PG+VG (Experimental): Subjects will then be instructed how to use the NFEC (eGo-T® with LED display) for 1 week of regularly vaping NFEC containing 50% PG and 50% VG. Subjects will be given the eGo-T®, which contains a 1.2 ml refillable cartridge and a 1100 milliamp hours (mAh) battery with an LED display to record the number of puffs. Subjects will be asked to puff 100x per day (equivalent to ~10-11 cigarettes) for 7 days. We will accept a vaping range of 80-120 times a day.
  Interventions: Other: PG+VG

INTERVENTIONS:
Other: Propylene Glycol — inhaled Propylene Glycol (PG) by vaporing
  Arms: vape NFEC containing 100% PG
Other: vegetable glycerin — inhaled vegetable glycerin (VG) by vaporing
  Arms: vape 100% vegetable glycerin -VG
Other: PG+VG — inhaled PG+VG by vaporing
  Arms: vape PG+VG

SUMMARY:
This aim will examine the acute and subacute exposures to electronic cigarette (EC) vapor generated from e-liquids without nicotine (NFEC) on life-time non smokers subjects by measuring changes in nasal ion transport and TGF-β levels. Nasal ion transport will be assessed by nasal potential difference (NPD). Tumor growth factor (TGF)-β levels (mRNA and protein by ELISA) will be assessed on nasal cells and lavages.

DETAILED DESCRIPTION:
The recent introduction of electronic cigarettes (ECs) to provide habitual smokers a source of nicotine without the need to inhale tobacco smoke is thought to reduce toxicity to airway epithelial cells. The use of ECs decreases use of traditional cigarettes diminishes nicotine withdrawal symptoms leads to opposite effects on exhaled NO levels compared to tobacco and may diminish stimulation of reward centers in the brain leading to less dependence due to the lack of other tobacco-derived chemicals. The manufacturers of ECs tout comparative safety as a reason to switch from traditional tobacco cigarettes to their products. However the dearth of data supporting this claim led the FDA to issue warning letters to these companies. For now, the World Health Organization recommends against EC use until ECs have been properly evaluated. On the other hand, the American Association of Public Health Physicians support the use of ECs as a means of "Harms Reduction" since ECs provide nicotine without the myriad of other toxic chemicals produced from burning tobacco. These recommendations are mostly due to theoretical considerations and expert opinion. Due to the novelty of the ECs, many concerns of their safety on health and long-term nicotine addiction remain unanswered due to a lack of studies that comprehensively evaluate their toxicity in the airways.

Moreover, ECs produce vapor mainly from propylene glycol (PG) or vegetable glycerin (VG) that are blended at different concentrations, making comprehensive testing more difficult.

The lack of consistent results demands a full evaluation of EC toxicity in the airway even when nicotine is not inhaled.

In our laboratory using cultures of primary normal human bronchial epithelial(NHBE) cells (either differentiating or fully differentiated) exposed to EC vapor or an equivalent volume of filtered air we have demonstrated that EC vapor can be delivered to fully differentiated NHBE cells and that high, but realistic puff numbers decrease ciliary beat frequency (CBF) as well as Large, Ca2+-activated K+ channels (BK channel) (the pore forming α subunit KCNMA1) and Forkhead box protein (FOXJ)-1 expression. We also have preliminary data of smoke exposure in vitro and in vivo, showing a negative effect of cigarette smoke and nicotine on parameters of mucociliary clearance (MCC) and nasal potential difference (NPD), a way to assess ion transport in vivo. These changes occurred in a TGF-β-dependent manner.

This study is designed to evaluate the airway toxicity of NFECs (Aim 2.1 of the project "Adverse effects of inhaled nicotine from tobacco and e-cigarettes").

PRIMARY ENDPOINT As the primary endpoint, we will assess the consequences of vaping EC liquid with no nicotine (NFEC) on cystic fibrosis transmembrane (CFTR)- and calcium-activated chloride channel (CaCC)-mediated chloride conductance in lifetime non-smokers using nasal potential difference (NPD) measurements.

We will use NPD as a primary endpoint because changes in most clinical parameters will only be seen after months or even years of exposure. For that particular reason, there is a recent surge to find alternative biomarkers that may be used as surrogate endpoints in shorter clinical trials. Since NPD directly measures the changes in ion transport expected to influence MCC and therefore overall outcome and since changes of NPD measurements are indirectly linked to lung function changes and MCC in trials with cystic fibrosis (CF) patients, we believe that NPD lends itself as a reasonable surrogate for MCC for this study.

SECONDARY ENDPOINTS Nasal nitric oxide and TGF-ß levels in nasal lavage and cells will be also collected to correlate with the changes on NPD results after exposure to NFEC.

STUDY DESIGN This aim will examine whether acute and subacute exposures to NFEC vapors have adverse effects on lifetime non-smokers by measuring changes in nasal ion transport and TGF-β levels. Nasal ion transport will be assessed by nasal potential difference (NPD), which measures the voltage potential resulting from epithelial ion fluxes (both Na+ absorption and Cl- and K+ secretion at the mucosal surface in vivo. In normal airway epithelia, Na+ absorption is the primary ion transport activity so that the resulting airway surface potential difference is negative with reference to the interstitium. Ion transport across nasal epithelia is representative for findings in distal airways. We also believe that NPD is a reasonably sensitive biomarker for this study as discussed below. Therefore, we will evaluate the acute effects of NFEC vapor generated from the nicotine-carrier system ("e-liquid" without nicotine) and the subacute effect after a 7-days exposure to the NFEC.

Since the major difference between the ECs is the amount of vapor produced per puff, we will focus on a commonly used mini and mid-sized EC: Halo (The Halo company, USA) and eGo-T® (Joyetech Co., Ltd., ShenZhen China), and examine different vapor fluids or "e-liquids" (100% PG, 50% PG/50% VG and 100% VG) without nicotine.

ELIGIBILITY:
Inclusion Criteria:

INCLUSION CRITERIA:

* Subjects will be over 18 years of age.
* Healthy life-time non-smokers

Exclusion Criteria:

* Presence of airflow obstruction (COPD, asthma, bronchiectasis)
* Other concomitant inflammatory pulmonary disorders
* Subjects with known pulmonary malignancies within 5 years
* Subjects with prior thoracic surgery
* Subjects with respiratory infection that required use of oral corticosteroids and/or antibiotics within the prior 3 months
* Subjects with allergies to study medications
* Subjects incapable of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-22 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
changes on nasal potential difference (NPD) measurements | before and after 7 days of vapor
  NPD will be measured at baseline and 7 days after the vapor

SECONDARY OUTCOMES:
changes on nasal nitric oxide | before and after 7 days of vapor
  Nitric oxide will be measured at baseline and 7 days after the vapor
changes on TGF-ß levels in nasal lavage | before and after 7 days of vapor
  TGF-ß will be measured at baseline and 7 days after the vapor

CONTACTS AND LOCATIONS:
Overall Officials: Michael Campos, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States